CLINICAL TRIAL: NCT06484348
Title: Deciphering the Interactions Between Food Intake, Sleepiness, and Nighttime Sleep Quality in Patients With Type 1 Narcolepsy and Idiopathic Hypersomnia
Acronym: NARCOFOOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL22_0943
Record Dates: First submitted 2024-05-27; First posted 2024-07-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Narcolepsy Type 1; Idiopathic Hypersomnia
Keywords: Narcolepsy type 1; Idiopathic Hypersomnia; Obesity; Food intake; Disrupted nighttime sleep
MeSH Terms: conditions — Idiopathic Hypersomnia; Obesity

STUDY DESIGN:
Intervention Model Description: A total of 20 NT1 patients, 20 IH patients and 20 Healthy Controls (HC) matched for age and gender will be prospectively included. The NT1 patients and HC groups will also matched for and be split into 2 subgroups of 10 participants according to BMI (<25 kg/m2 and ≥ 25 kg/m2). IH will be matched to NT1 for wake-promoting drugs dosage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NT1 (Experimental): Patients with Narcolepsy type 1 will be included in this arm.
  They will have following interventions :
  1. monitoring of eating behaviors (meals' photos) and sugar consumption (FreeStylePro sensor measuring interstitial glucose)
  2. monitoring of sleep/wake rhythm (diary and actigraphy)
  3. monitoring of nocturnal sleep parameters (Somfit device)
  4. monitoring of sleepiness (Karolinska sleepiness scale and EEG markers of sleepiness with the Somfit device) before and after meals
  Interventions: Behavioral: Monitoring of eating behaviors; Behavioral: Monitoring of sleep/wake rhythm; Behavioral: Measure of nocturnal sleep parameters; Behavioral: Measure of sleepiness
- IH (Active Comparator): Patients with Idiopathic Hypersomnia will be included in this arm.
  They will have following interventions :
  1. monitoring of eating behaviors (meals' photos) and sugar consumption (FreeStylePro sensor measuring interstitial glucose)
  2. monitoring of sleep/wake rhythm (diary and actigraphy)
  3. monitoring of nocturnal sleep parameters (Somfit device)
  4. monitoring of sleepiness (Karolinska sleepiness scale and EEG markers of sleepiness with the Somfit device) before and after meals
  Interventions: Behavioral: Monitoring of eating behaviors; Behavioral: Monitoring of sleep/wake rhythm; Behavioral: Measure of nocturnal sleep parameters; Behavioral: Measure of sleepiness
- HC (Active Comparator): Healthy Controls will be included in this arm.
  They will have following interventions :
  1. monitoring of eating behaviors (meals' photos) and sugar consumption (FreeStylePro sensor measuring interstitial glucose)
  2. monitoring of sleep/wake rhythm (diary and actigraphy)
  3. monitoring of nocturnal sleep parameters (Somfit device)
  4. monitoring of sleepiness (Karolinska sleepiness scale and EEG markers of sleepiness with the Somfit device) before and after meals
  Interventions: Behavioral: Monitoring of eating behaviors; Behavioral: Monitoring of sleep/wake rhythm; Behavioral: Measure of nocturnal sleep parameters; Behavioral: Measure of sleepiness

INTERVENTIONS:
Behavioral: Monitoring of eating behaviors — Overall eating behaviors will be assessed from pictures of consumed food and drinks taken by the participants with their smartphones. A complete assessment of eating habits will be carried out daily for 4 days. For each photo, the participants will indicate the reasons why they ate by completing analogical scales (hunger, craving, sleepiness, stress, negative emotion) and an open question (other reason). These data will be used to determine the reason and timing of food intake and the number of calories ingested for each food category. Eating behaviors specifically related to sugar intake will be monitored using the FREESTYLE PRO® sensor. This small device is used routinely for diabetes care and is placed on the back of the arm. The system is designed to measure glucose levels in the interstitial fluid every 15 minutes for up to 14 days. The recorded data can be downloaded by an investigator using the FREESTYLE LIBRE PRO® reader.
Behavioral: Monitoring of sleep/wake rhythm — The sleep-wake rhythm will be measured continuously during the 5 days, both subjectively (sleep diary) and objectively, using the GT9X "LINK" ACTIGRAPH.
Behavioral: Measure of nocturnal sleep parameters — The quality and quantity of the participants' sleep will be recorded using the SOMFIT® device. This non-invasive portable device will allow the determination of sleep architecture as well as sleep EEG microstructure.
Behavioral: Measure of sleepiness — Sleepiness will be assessed by the Karolinska Sleepiness Scale (KSS) at the initiation of food intake and 30 min and 2 hours afterwards, and by analysis of EEG activity recorded by the SOMFIT® over a time window surrounding food intake. Indeed, participants will also be asked to wear the device as much as possible during the day when they are at home in order to explore sleepiness markers during wakefulness.

SUMMARY:
Links between sleep and food intake are manyfold. In healthy individuals, sleep deprivation promotes obesity by stimulating food intake of high glycemic index (GI) foods. Conversely, high GI foods induce sleepiness. Obesity is observed in 30-50% of patients with Narcolepsy type 1 (NT1). Its determinism may involve transient changes in basal metabolism at the early stage of the disease, eating disorders, disrupted nighttime sleep and sleepiness. In contrast, patients suffering from idiopathic hypersomnia (IH), whose nocturnal sleep is generally long and of good quality, rarely present with obesity. By studying the relationships between diet, body composition and sleep patterns in these two populations and in healthy controls, the NARCOFOOD study aims to provide a better understanding of the determinants of obesity in narcolepsy and, more generally, of the effects of food intake on sleepiness.

Patients will be recruited at the Lyon and Clermont-Ferrand sleep centers and Controls at the Lyon Neuroscience Research Center. Data from clinical evaluation (including body mass index and body composition), and questionnaires (sleep quality, insomnia, sleepiness, anxiety and depression, impulsivity, eating behaviors) will be collected. During 4 days, at home, the following parameters will be explored : 1) eating behaviors (meals' photos) and sugar consumption (FreeStylePro sensor measuring interstitial glucose) 2) sleep/wake rhythm (diary and actigraphy) 3) nocturnal sleep parameters (Somfit device) 4) sleepiness (Karolinska sleepiness scale and EEG markers of sleepiness with the Somfit device) before and after meals.

The hypothesis is that increased sleepiness would favor food intake of high GI foods, which would worsen sleepiness in all 3 groups, with a more pronounced effect in NT1. Compared to IH patients and controls, NT1 patients may present more snacking of high GI foods, especially at night if sleep is disrupted, and this would be correlated with body composition.

The findings will help to better understand the mechanisms of obesity in narcolepsy and may lay the ground for the development of new therapeutic strategies in disorders of hypersomnolence, targeting dietary behaviors.

ELIGIBILITY:
Inclusion Criteria :

* Patients with NT1 or IH (ICSD-3-TR) or Healthy Controls without sleep disorder
* Familiar use of a smartphone

Exclusion Criteria :

* Untreated moderate or severe sleep apnea syndrome;
* Cognitive disorders incompatible with the protocol;
* Unstable treatment or treatment with sodium oxybate;
* Unstable medical or psychiatric pathology;
* Shift work;
* Pregnancy or breastfeeding;
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
impact of glycaemic load on sleepiness 2 hours after lunch | 2 hours after lunch, from day 1 to day 3
  To compare the impact of glycaemic load on sleepiness assessed by the Karolinska sleepiness scale (KSS) 2 hours after lunch (midday meal or food intake between 11 a.m. and 4 p.m.) between the 3 groups of participants (NT1, IH, CT).
  Correlation coefficient between the quantitative measure of glycaemic load assessed by the area under the interstitial glucose curve for 2 hours after the start of lunch and the change in sleepiness assessed by the variation in the score on the KSS between the pre- and post-prandial period, with post-prandial assessment 2 hours after the start of lunch.

SECONDARY OUTCOMES:
impact of glycaemic load on sleepiness 2 hours after the start of each food intake | 2 hours after the start of each food intake, from day 1 to day 3
  To compare the impact of glycaemic load on sleepiness assessed by the KSS 2 hours after the start of each food intake (breakfast + lunch + dinner + snacks) between the 3 groups of subjects (NT1, IH, CT).
  Correlation coefficient between the quantitative measure of glycaemic load assessed by the area under the interstitial glucose curve for 2 hours after the start of each food intake (breakfast + lunch + dinner + snacks) and the change in sleepiness assessed by the change in score on the KSS instantaneous sleepiness scale between the pre- and post-prandial periods, with post-prandial assessment 2 hours after the start of each food intake (breakfast + lunch + dinner + snacks).
impact of glycaemic load on sleepiness 30 min after the start of lunch and each food intake | 30 min after the start of lunch and each food intake, from day 1 to day 3
  To compare the impact of glycaemic load on sleepiness assessed by the KSS 30 min after the start of lunch and each food intake (breakfast + lunch + dinner + snacks) between the 3 groups of subjects (NT1, IH, CT).
  Correlation coefficient between the quantitative measure of glycaemic load assessed by the area under the interstitial glucose curve for 30min after the start of lunch alone and after all meals (breakfast + lunch + dinner + snacks) and the change in sleepiness assessed by the variation in the score on the KSS instantaneous sleepiness scale between the pre- and post-prandial periods ((post-pre)/pre), with postprandial assessment 30min after the start of lunch or of all food intake (breakfast + lunch + dinner + snacks).
impact of food intake on sleepiness 30 minutes and 2 hours after the start of lunch and each food intake | 30 minutes and 2 hours after the start of lunch and each food intake, from day 1 to day 3
  To compare the impact of food intake (total calorie intake, fat intake, protein intake) on sleepiness assessed by the KSS 30 minutes and 2 hours after the start of lunch and each food intake (breakfast + lunch + dinner + snacks) between the 3 groups of subjects (NT1, IH, CT).
  Correlation coefficient between the measurement of total calorie intake, fat intake, protein intake, carbohydrate intake weighted by the glycaemic index associated with food intake and the change in sleepiness assessed by the variation in the score on the KSS instantaneous sleepiness scale between the pre- and post-prandial periods, with postprandial assessment 30 minutes and 2 hours after the start of lunch or of all food intake (breakfast + lunch + dinner + snacks).
impact of glycaemic load and food intake on sleepiness 30 minutes and 2 hours after the start of lunch and each food intake | 30 minutes and 2 hours after the start of of lunch and each food intake, from day 1 to day 3
  To compare the impact of glycaemic load and food intake (total calorie intake, lipids intake, proteins intake) on motor activity 30 minutes and 2 hours after the start of lunch and each food intake (breakfast + lunch + dinner + snacks) between the 3 groups. Motor activity will be measured by actigraphy (time spent with motor activity lower than the average motor activity recorded while awake over 4 days) within 30 minutes and between 30 minutes and 2 hours after the start of food intake.
  Correlation coefficient between the measurement of glycaemic load assessed by the area under the interstitial glucose curve, total calorie intake, fat intake, protein intake, carbohydrate intake weighted by the glycaemic index associated with food intake and motor activity measured by actimetry (time spent with motor activity less than the average motor activity recorded awake over 4 days) within 30 minutes and in the period 30 minutes - 2 hours after the start of food intake.
Impact of glycaemic load and food intake on EEG markers of sleepiness 30 minutes and 2 hours after the start of lunch and each food intake | 30 minutes and 2 hours after the start of lunch and each food intake, from day 1 to day 3
  To compare the impact of glycaemic load and food intake (total calorie intake, lipids, proteins, carbohydrates) on EEG markers of sleepiness 30 minutes and 2 hours after the start of lunch and each food intake (breakfast + lunch + dinner + snacks) between the 3 groups of subjects (NT1, IH, CT).
  Correlation coefficient between the measurement of glycaemic load assessed by the area under the interstitial glucose curve, total calorie intake, fat intake, protein intake, carbohydrate intake weighted by the glycaemic index associated with food intake and the presence of EEG sleepiness markers (slow wave index (n/min), delta power (relative to the mean delta power during the previous day), cumulative number and duration of sleep and microsleep episodes) assessed by the SOMFIT® device within 30 minutes and between 30 minutes and 2 hours after the start of food intake.
Impact of subjective and objective markers of sleepiness on food intake | During all food intakes, from day 1 to day 3
  To compare the impact of subjective and objective markers of sleepiness on food intake during lunch alone and during all food intakes between the 3 groups.
  Correlation coefficient between food intake (total calorie intake, fat, protein and carbohydrate intake weighted by the glycaemic index for each food intake, area under the interstitial glucose curve) for lunch alone and for all food intakes in the 3 groups and (1) the score on the KSS instantaneous sleepiness scale (10 min) before each food intake; (2) motor activity measured by actimetry in the hour before each food intake (time spent with motor activity greater than the average motor activity recorded during the previous 4 days); (3) EEG markers of sleepiness in the hour before each food intake (slow wave index, delta power in the hour before each food intake, number and cumulative duration of sleep and microsleep episodes).
relationship between the temporal course of interstitial glucose and that of objective markers of sleepiness | from 1 hour before to 2 hours after each food intake, from day 1 to day 3
  To compare the relationship between the temporal course of interstitial glucose and that of objective markers of sleepiness (actigraphy and EEG) measured in the period from 1h before to 2h after lunch and each food intake (breakfast + lunch + dinner + snacks) between the 3 groups of subjects (NT1, IH, CT).
  2 to 2 cross-correlations between the temporal evolution of interstitial glucose levels, spectral power in the delta band of the EEG (SOMFIT ®), and the number of movements recorded by actigraphy averaged every 5 minutes from t=-60min to t=120min in relation to the start of lunch alone and each food intake (breakfast + lunch + dinner + snacks). The maximum power of the correlation and the time lag for which the correlation is maximum will be compared between the 3 groups of subjects (NT1, IH, CT). A more detailed analysis will also be carried out on all subjects and food intakes using temporal auto-regressive networks.
To compare the distribution (time, night versus day) of food intake between the 3 groups. | From day 1 to day 3
  Distribution (times, % night (after bedtime) versus day (after waking)) of food intake in the 3 groups during the observation period.
To compare the motivation for eating between the 3 groups. | From day 1 to day 3
  Subjective motives (habit, hunger, desire to eat, stress, hypovigilance) of food intake in the 3 groups assessed by questionnaires before food intake during the observation period.
  This will be measured previous to each food intake by several questions evaluating the reason for food intake: 1) Habits (is it one of your usual meal ? yes/no) 2) Hunger (Are you hungry ?) 3) What is your desire to eat right now ? 4) Do you feel stressed or anxious ? 5) KSS
To compare the quantity of food intake between the 3 groups. | From day 1 to day 3
  Quantity (total calorie intake) of food intake in the 3 groups during the observation period.
To compare the quality of food intake between the 3 groups. | From day 1 to day 3
  Quality (fat, protein, carbohydrate intake weighted by glycaemic index, area under the interstitial glucose curve) of food intake in the 3 groups during the observation period. This will be assessed 1) by pictures taken by the participants before and after each meal: the pictures will be evaluated by a professional dietician used to doing quantifications of food composition based on such pictures 2) by the area under the interstitial glucose curve obtained with the FreeStyle Pro device, during the 30 min and 2h following the meal
links between the characteristics of food intake and indicators of overweight/obesity, sleepiness and sleep quality | At baseline and from day 1 to day 3
  To explore the links between the characteristics of food intake (distribution, quality, quantity) and indicators of overweight/obesity (BMI, % body fat), sleepiness (ESS) and sleep quality (measured by SOMFIT®) in all subjects and to compare them between the 3 groups of subjects (NT1, IH, CT).
  Correlation between the mean characteristics over the observation period of food intake (distribution: schedules, % night versus day; quantity: total caloric intake; and quality: fat, protein, carbohydrate intake weighted by glycaemic index, area under the interstitial glucose curve) and (1) BMI and (2) body composition (% fat mass and lean mass measured by impedancemetry) at inclusion in the 3 groups (3) sleepiness (ESS at baseline) (4) quality of sleep at night (sleep efficiency measured by SOMFIT®).
Identify the factors associated with the presence of eating disorders | At baseline
  Identify the factors associated with the presence of eating disorders (assessed by the Eating Disorder Examination Questionnaire (EDEQ)-6) in all subjects and compare them between the 3 groups.
  The factors explored will be: age, sex, BMI, body composition, diagnostic category (and disease severity), medications, anxiety/depression, sleepiness, presence of parasomnias, presence/severity of restless legs syndrome, insomnia severity, apathy, impulsivity, alexithymia, sedentary, chronotype, night-time sleep efficiency using actigraphy and SOMFIT®.
Identification of factors associated with the presence of binge eating behaviors | At baseline and from day 1 to day 3
  Identify the factors associated with the presence of binge eating behaviors (assessed by the BES) in all subjects and compare them between the 3 groups.
  The factors explored will be: age, sex, BMI, body composition, diagnostic category (and disease severity), medications, anxiety/depression, sleepiness, presence of parasomnias, presence/severity of restless legs syndrome, insomnia severity, apathy, impulsivity, alexithymia, sedentary, chronotype, night-time sleep efficiency using actigraphy and SOMFIT®.
Identification of factors associated with the presence of night eating syndrome | At baseline and from day 1 to day 3
  Identify the factors associated with the presence of night eating syndrome (assessed by the NEQ) in all subjects and compare them between the 3 groups.
  The factors explored will be: age, sex, BMI, body composition, diagnostic category (and disease severity), medications, anxiety/depression, sleepiness, presence of parasomnias, presence/severity of restless legs syndrome, insomnia severity, apathy, impulsivity, alexithymia, sedentary, chronotype, night-time sleep efficiency using actigraphy and SOMFIT®.
Identification of factors associated with the characteristics of eating behaviors | At baseline and from day 1 to day 3
  Identify the factors associated with the characteristics of eating behaviors (assessed by the distribution, quantity and quality of food intake) in all subjects and compare them between the 3 groups.
  The factors explored will be: age, sex, BMI, body composition, diagnostic category (and disease severity), medications, anxiety/depression, sleepiness, presence of parasomnias, presence/severity of restless legs syndrome, insomnia severity, apathy, impulsivity, alexithymia, sedentary, chronotype, night-time sleep efficiency using actigraphy and SOMFIT®.
response of interstitial glycaemia levels following a calibrated glucose load test and the impact of this response on subjective and objective markers of sleepiness | from t0 to t120 minutes after a calibrated glucose load, at the end of the study (between day 4 and day 7)
  To compare the response of interstitial glycaemia levels following a calibrated glucose load test and the impact of this response on subjective and objective markers of sleepiness using cross-correlations between the time courses of these variables during the 2 hours following glucose intake between the 3 groups.
  Area under the interstitial glucose curve from t0 to t120 minutes, maximum value reached, timing of maximum, and slope of decrease in glucose levels after maximum value will be compared between the 3 groups.
  Coefficient of 2 to 2 cross-correlations between the temporal evolution of interstitial glucose levels, the drowsiness score assessed by the KSS scale, the number of movements recorded by actimetry and the spectral power in the delta band of the EEG averaged every 15 minutes for 2 hours following ingestion of a calibrated glucose load. The maximum power of the correlation and the time lag at which the correlation is maximal will be compared between the 3 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Laure PETER-DEREX, MD-PhD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Unité de Neurophysiologie-sommeil, Département de Neurologie, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Center for Sleep Medicine, Hospices Civils de Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No